CLINICAL TRIAL: NCT06496880
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Group Study to Evaluate Efficacy of OxyjunTM on Cardiac Pumping Capacity as Well as Work Productivity in Individuals With Metabolic Risk
Brief Title: A Study to Evaluate the Efficacy of OxyjunTM on Cardiac Pumping Capacity as Well as Work Productivity in Individuals With Metabolic Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/240301/OXY/CPC
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Disorder
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Placebo-controlled, Parallel Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OxyjunTM (Active Comparator): One capsule daily to be taken after breakfast for 56 days
  Interventions: Dietary Supplement: Oxyjun TM
- Microcrystalline Cellulose (Placebo Comparator): One capsule daily to be taken after breakfast for 56 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oxyjun TM — One capsule daily to be taken after breakfast for 56 days
  Arms: OxyjunTM
Dietary Supplement: Placebo — One capsule daily to be taken after breakfast for 56 days
  Arms: Microcrystalline Cellulose

SUMMARY:
A Randomized, Double Blind, Placebo-controlled, Parallel Group Study to Evaluate Efficacy of OxyjunTM on Cardiac Pumping Capacity as well as Work Productivity in Individuals with Metabolic Risk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either sex, aged more than equal to 45 to less than equal to 70 years at the time of screening with BMI more than equal to 25 kg/metre square to less than equal to 34.9 kg/metre square.
* Individuals with normal to high blood pressure (BP) [systolic BP more than equal to 120 mmHg and less than equal to 159 mmHg and/or diastolic BP more than equal to 80 mmHg and less than equal to 89 mmHg].
* Individuals with waist circumference more than equal to 40 inches for men or 35 inches for women.
* Individuals with normal to mildly deranged 'Left ventricular ejection' as per American College of Cardiology: LVEF more than equal to 45% and less than equal to 55%.
* Fasting glucose level of more than equal to 110 mg/dL and less than equal to 160 mg/dL (without medication or with maximum 500 mg of daily dose of Metformin).
* Individuals with Aspartate aminotransaminase (AST) and Alanine transaminase (ALT) within 2 times upper normal limit (ULN).
* Individuals with 1.5 x Upper Normal Limit (ULN) of Creatinine.
* Individuals having following values of haemoglobin:

  1. Female - more than equal to 11 mg/dl
  2. Male - more than equal to 12 mg/dl
* Individuals with thyroid stimulating hormone (TSH) levels in between 0.27 IU/ml and 5 IU/ml both values included.
* Individuals who demonstrate their willingness to participate in the study and comply with the study procedures and required visits.
* Willing to abstain from caffeine for 12 hours prior to the visit
* Willing to abstain from alcohol and related products consumption for 48 hours prior to study visits
* Must be literate, having the ability to understand, complete the study-based questionnaires, requirements and sign a written informed consent form, which must be completed prior to study specific requirements being performed.

Exclusion Criteria:

* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgement of the investigator, would interfere with the individuals ability to provide informed consent, comply with the study protocol, or put the individual at undue risk.
* Using Omega fish oil supplements, anticonvulsants, Coenzyme Q10, Vitamin K2, proton pump inhibitors, loop diuretics, anticoagulants, barbiturates, anti-epileptic medications and any herbal supplements (e.g. flax seeds, chia seeds).
* Chronic use of anti-inflammatory medications (more than equal to 5 tablets/20 days in last 3 months).
* Individuals having a history of smoking or currently smoking or using any form of smokeless tobacco.
* High-risk drinking as defined by consumption of 4 or more drinks of alcohol containing beverages on any day or 10 or more drinks of alcohol containing beverages per week for women and 5 or more drinks of alcohol containing beverages on any day or 14 or more drinks of alcohol containing beverages per week for men.
* Individuals unable to walk. Individuals with a history of chronic caffeine use with more than 3 cups of caffeinated beverage/ day.
* Individuals who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put him/her at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.
* Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
* Females undergoing hormone replacement treatments.
* Peri- or post-menopausal females having less than equal to 1 year of irregular or complete absence of menstrual cycle.
* Those unwilling to abstain from other dietary supplements or medication (e.g. Hepatoprotective agents and complementary and alternative medicine).
* Have participated in a study of an investigational product 90 days prior to the screening.
* Individuals with known or suspected hypersensitivity or intolerance to Investigational product.
* Individuals who are unable to comply with study requirements.
* Individuals with a history of autoimmune disorders
* Individuals with a history of immunocompromised status
* Any clinical signs or symptoms that in the opinion of the investigator can jeopardize the outcome of the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of 8-week oral consumption of OxyjunTM on left ventricular function as evaluated by Left ventricle ejection fraction (LVEF). | Screening
  LVEF is the fraction of chamber volume ejected during systole (stroke volume or SV) in relation to the volume of blood in the ventricle at the end of diastole (end-diastolic volume or EDV). The LVEF will be assessed by using M-mode 2D Echo.
  LVEF is calculated using the formula- LVEF: [SV/EDV] x 100
To evaluate the effect of 8-week oral consumption of OxyjunTM on left ventricular function as evaluated by Left ventricle ejection fraction (LVEF). | Day 28
  LVEF is the fraction of chamber volume ejected during systole (stroke volume or SV) in relation to the volume of blood in the ventricle at the end of diastole (end-diastolic volume or EDV). The LVEF will be assessed by using M-mode 2D Echo.
  LVEF is calculated using the formula- LVEF: [SV/EDV] x 100
To evaluate the effect of 8-week oral consumption of OxyjunTM on left ventricular function as evaluated by Left ventricle ejection fraction (LVEF). | Day 56
  LVEF is the fraction of chamber volume ejected during systole (stroke volume or SV) in relation to the volume of blood in the ventricle at the end of diastole (end-diastolic volume or EDV). The LVEF will be assessed by using M-mode 2D Echo.
  LVEF is calculated using the formula- LVEF: [SV/EDV] x 100

SECONDARY OUTCOMES:
To evaluate the effect of 8-week oral consumption of Oxyjun TM on Cardiac pumping capacity as evaluated by the ventricular stroke volume and cardiac output. | Screening, Day 28 and Day 56
  Cardiac output is determined by multiplying heart rate and stroke volume and is typically measured in liters per minute cardiac output is expressed as CO = HR × SV.
  The normal range for stroke volume is typically 55-100 mL. An average resting heart rate is approximately 75 beats per minute (bpm), but it can vary between 60-100 bpm in some individuals.
  The normal cardiac output falls within the range of 4.0-6.0 L/min at rest
To evaluate the effect of 8-week oral consumption of Oxyjun TM on Responder to the product as assessed by the number of the participant having LVEF more than equal to 5 units increase. | Screening, Day 28 and Day 56
  Echocardiography define normal left ventricular ejection fraction (LVEF) as greater than 50% and greater than 55%, respectively.
To evaluate the effect of 8-week oral consumption of OxyjunTM on Work Productivity as assessed by the Work Productivity and Activity Impairment Questionnaire | Day 0, Day 28 and Day 56
  The Work Productivity and Activity Impairment (WPAI) questionnaire stands as a thoroughly validated tool designed to assess impairments in both work-related tasks and general activities.
  In this study, a 10 point Visual Analogue scale is used to evaluate how health problems affect the participant's ability to do their regular activity where 0 means no effect and 10 means complete hinderance in daily activities.
To evaluate the effect of 8-week oral consumption of Oxyjun TM on Cardiac risk as assessed by the N-terminal pro b-type natriuretic peptide (NT-Pro BNP) | Day 0 and Day 56
  NT-Pro BNP levels have been noted in various cardiovascular conditions, encompassing chronic heart failure and left ventricular dysfunction.
  Normal reference range considered in this study for males and females for NT-Pro BNP is <125 pg/ml
To evaluate the effect of 8-week oral consumption of Oxyjun TM on Physical activity as assessed by IPAQ-SF questionnaire | Day 0, day 28 and day 56
  The IPAQ-SF is a standardized and culturally adaptable tool to assess habitual physical activity in individuals across the globe.
  Scoring a HIGH level of physical activity on the IPAQ-SF means the physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ-SF means one is doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ-SF means that the participant is not meeting any of the criteria for either MODERATE or HIGH levels of physical activity.

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Sigma Hospital, Mumbai, Maharashtra
  - Vedant Multispeciality Hospital, Pune, Maharashtra
  - Umarji Mother & Child Care Hospital, Pune, Maharashtra
  - Swara Hospital, Thane, Maharashtra
  - Silver Birch Multispecialty Hospital, Pune, Maharshtra
  - Upendra Medicare Hospital, Varanasi, Uttar Pradesh
  - Janta hospital & Maternity Centre, Varanasi, Uttar Pradesh